CLINICAL TRIAL: NCT05134233
Title: Investigation of Low-intensity Focused Ultrasound Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-882
Record Dates: First submitted 2021-11-10; First posted 2021-11-24 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Development of LIFU for Clinical Purposes
Keywords: low-intensity focused ultrasound; transcranial magnetic stimulation

STUDY DESIGN:
Intervention Model Description: Multi-visit study, testing various LIFU parameters per session
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parameter Trials (Experimental): Approximately 36 parameter combinations will be tested per study session, expected 6 sessions of trials. Response recorded using TMS and EMG.
  Interventions: Device: Low-intensity Focused Ultrasound

INTERVENTIONS:
Device: Low-intensity Focused Ultrasound — LIFU application using various parameters, responses of neuromodulation recorded using TMS and EMG.

SUMMARY:
This project examines the effects of different brain stimulation settings on muscle contractions. The investigators believe this study will help to better understand noninvasive brain stimulation techniques that may have the potential to aid in addiction, pain, and mental health issues. Participants undergo structural imaging, an fMRI and CT. These images are used to align the low-intensity focused ultrasound (LIFU) and transcranial magnetic stimulation (TMS) devices to temporarily change brain activity. Electromyography (EMG) will be used to record muscle contractions on the hand.

ELIGIBILITY:
Inclusion Criteria:

* Above criteria and must understand and speak English.

Exclusion Criteria:

* Contraindications to MRI, CT, or TMS

  1. Claustrophobia
  2. Pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
  3. Pregnancy
  4. Active medical disorder or treatment with potential CNS effects
  5. History of neurologic disorder
  6. History of head injury resulting in loss of consciousness for >10 minutes
  7. History of alcohol or drug dependence
  8. Failure to provide a social security number or tax ID number. This is required for tax purposes or payment cannot be processed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legon W, Bansal P, Tyshynsky R, Ai L, Mueller JK. Transcranial focused ultrasound neuromodulation of the human primary motor cortex. Sci Rep. 2018 Jul 3;8(1):10007. doi: 10.1038/s41598-018-28320-1. PMID 29968768
- [Background] Fomenko A, Chen KS, Nankoo JF, Saravanamuttu J, Wang Y, El-Baba M, Xia X, Seerala SS, Hynynen K, Lozano AM, Chen R. Systematic examination of low-intensity ultrasound parameters on human motor cortex excitability and behavior. Elife. 2020 Nov 25;9:e54497. doi: 10.7554/eLife.54497. PMID 33236981
- [Background] Xia X, Fomenko A, Nankoo JF, Zeng K, Wang Y, Zhang J, Lozano AM, Chen R. Time course of the effects of low-intensity transcranial ultrasound on the excitability of ipsilateral and contralateral human primary motor cortex. Neuroimage. 2021 Nov;243:118557. doi: 10.1016/j.neuroimage.2021.118557. Epub 2021 Sep 4. PMID 34487826

RESULTS

PARTICIPANT FLOW:
Groups:
- Parameter Trials: Up to 15 parameter combinations will be tested per study session, expected up to 6 sessions of trials. Response recorded using TMS and EMG.
  Low-intensity Focused Ultrasound: LIFU application using various parameters, responses of neuromodulation recorded using TMS and EMG.
Period: Overall Study
Arm/Group | Parameter Trials
Started | 23
Completed | 19
Not Completed | 4
Not completed — Pregnancy | 1
Not completed — MEP value too low | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Parameter Trials
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 29 [20 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Waveforms
Description: Changes in waveform peak will be observed per each variable application of LIFU
Time Frame: Outcome measured throughout study participation - an average of 4 weeks per participant.
Population: One participant data set had artifacts that could not be removed while leaving usable MEP data.
Measure: Mean (Standard Deviation); unit: percentage of baseline MEP mV
Arm/Group | Parameter Trials
Number analyzed (Participants) | 18
percentage of baseline MEP mV
  Parameter 1 (6W/cm2-1%DC-100msec) | 1.06 (0.12)
  Parameter 2 (6W/cm2-10%DC-100msec) | 1.10 (0.12)
  Parameter 3 (6W/cm2-30%DC-100msec) | 0.97 (.10)
  Parameter 4 (6W/cm2-50%DC-100msec) | 0.99 (0.10)
  Parameter 5 (6W/cm2-70%DC-100msec) | 1.03 (0.13)
  Parameter 6 (6W/cm2-1%DC-500msec) | 0.80 (0.10)
  Parameter 7 (6W/cm2-10%DC-500msec) | 0.84 (0.10)
  Parameter 8 (6W/cm2-30%DC-500msec) | 0.70 (0.08)
  Parameter 9 (6W/cm2-50%DC-500msec) | 0.81 (0.11)
  Parameter 10 (6W/cm2-70%DC-500msec) | 0.75 (0.08)
  Parameter 11 (24W/cm2-1%DC-100msec) | 0.86 (0.09)
  Parameter 12 (24W/cm2-10%DC-100msec) | 0.93 (0.11)
  Parameter 13 (24W/cm2-30%DC-100msec) | 1.01 (0.12)
  Parameter 14 (24W/cm2-50%DC-100msec) | 0.91 (0.12)
  Parameter 15 (24W/cm2-70%DC-100msec) | 0.91 (0.09)
  Parameter 16 (24W/cm2-1%DC-500msec) | 0.75 (0.07)
  Parameter 17 (24W/cm2-10%DC-500msec) | 0.79 (0.10)
  Parameter 18 (24W/cm2-30%DC-500msec) | 0.84 (0.10)
  Parameter 19 (24W/cm2-50%DC-500msec) | 0.93 (0.13)
  Parameter 20 (24W/cm2-70%DC-500msec) | 0.84 (0.09)
  Parameter 21 (continuous- 6W/cm2-35000 cycles) | 0.84 (.11)
  Parameter 22 (continuous- 24W/cm2-35000 cycles) | 1.05 (0.13)
  Parameter 23 (continuous- 6W/cm2-75000 cycles) | 1.10 (0.13)
  Parameter 24 (continuous- 24W/cm2-75000 cycles) | 0.99 (0.10)

ADVERSE EVENTS:
Time Frame: Beginning (prior to study tasks) and end of each study visit, visits occurring over an average of 4 weeks - participants completed report of symptoms questionnaire.
Description: Collected a Report of Symptoms Questionnaire pre/post LIFU application at each study visit.
Arm/Group | Parameter Trials
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT05134233/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT05134233/SAP_001.pdf